CLINICAL TRIAL: NCT03694054
Title: Exploratory Evaluation of Family Caregiver Application (FCA) on Quality Among Persons With Lung Cancer and Their Family Caregivers
Brief Title: Care Coordination in Oncology, Quality Among Patients With Lung Cancer and Their Caregivers
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Geisinger Clinic (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2018-0172
Record Dates: First submitted 2018-09-11; First posted 2018-10-03 (Actual); Last update posted 2019-04-09 (Actual); Status verified 2019-04

CONDITIONS: Lung Cancer
Keywords: Care Coordination; Oncology Care; Lung Cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Care coordination patients, caregivers (Experimental): Patients and caregivers enroll in using care coordination tool during oncology care and treatment.
  Interventions: Other: Care coordination tool
- Standard of care patients, caregivers (No Intervention): Patients and caregivers receive oncology care and treatment.
- Oncology Care Providers (Experimental): Oncology care providers with patients enrolled in care coordination tool.
  Interventions: Other: Care coordination tool

INTERVENTIONS:
Other: Care coordination tool — Participants will be asked to enroll in the care coordination tool, a health information technology solution that integrates cross-sector data to enhance communication and improve quality of care and performance outcomes. Patients will also be asked to provide consent to allow the study team to access additional health information via the electronic health record.
  Arms: Care coordination patients, caregivers; Oncology Care Providers

SUMMARY:
The Oncology Care Coordination study is designed to evaluate use of a care coordination tool for lung cancer patients and their caregiver on quality of care and performance outcomes. Eligible patients need to be receiving treatment at Geisinger. Participation in the study involves completion of surveys, permission to review information from the patient's electronic health record, and for some enrollment in the care coordination tool called Harmonized Care. Geisinger oncology care providers who have patients enrolled the study will be invited for interviews.

DETAILED DESCRIPTION:
The case-matched controlled design, exploratory evaluation study will look at how exposure to a care coordination tool impacts quality and performance indicators associated with oncology care from the perspective of patients, caregivers, and providers.

Geisinger research staff will recruit lung cancer patients and their caregivers across three Geisinger locations: Geisinger Medical Center (GMC), Geisinger Wyoming Valley Medical Center (GWV) and Geisinger Community Medical Center (GCMC). GMC will serve as the intervention site and GWV and GCMC as control sites.

Eligible participants will be identified by the study staff through the electronic health record as well as through clinical staff and approached in the oncology clinic as part of a schedule office visit and/or treatment. For the purpose of study awareness, informational flyers will be available to patients in the exam rooms, waiting rooms, and through Oncology Care's Multi-Disciplinary clinic. Participants will asked to identify a caregiver who will participate in the study as well, however this is not required.

Case dyads enrolled at the intervention site (GMC) will be asked to complete a survey when they join the study and at the end of the study. Participants will also be asked to enroll in the care coordination tool, a health information solution that integrates the patient, caregiver, and clinical data to enhance communication and improve quality of care and performance outcomes. Patients will also be asked to give permission to the study team to access their health information via the e electronic health record. Participants will be in the research study for about 8-10 weeks.

Control dyads enrolled at the control site (GWV and GCMC) will be asked to complete a survey eight weeks after consenting to participate. Patients will be asked to give permission to the study team to access their health information via the electronic health record. Participants will be in the research study for about 8-10 weeks.

The study will also enroll oncology care providers within the Medical Oncology or Radiation Oncology departments at GMC and who have patients enrolled in the study. Providers will be asked to participate in a 30-minute interview to get their feedback and insights on the care coordination tool.

ELIGIBILITY:
Inclusion Criteria:

Patients:

* Patients who are 18 years of age or older and diagnosed with lung cancer who 1) are scheduled to start Oncology Care (chemo and/or radiation-therapies) OR 2) on active Oncology Care and recently started within 3 weeks (<27 days for experimental arm; <56 days control arm)
* Receive care at GMC, GWV, or GCMC
* English-speaking
* Established/intends to establish a MyGeisinger Account (cases only)

Caregivers:

* Recognized/intends to be recognized as proxy for patient's MyGeisinger Account (cases only)
* English-speaking

Providers:

- Any health care provider within Medical Oncology or Radiation Oncology at GMC, where care coordination tool is standard of care, who has a patient enrolled.

Exclusion Criteria:

Patients:

* Patients who are not diagnosed with lung cancer.
* Patients who are diagnosed with lung cancer and are on active Oncology Care exceeding 3 weeks (>27 days experimental arm; >56 days control arm).

Providers:

* Any healthcare provider not within the Medical Oncology or Radiation Oncology departments.
* Any healthcare provider within Medical Oncology or Radiation Oncology who does not have a patient enrolled (Case Dyad).

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2018-06-04 (Actual); Primary Completion 2019-02-28 (Actual); Study Completion 2019-03-31 (Actual)

PRIMARY OUTCOMES:
Patient Satisfaction | 8 weeks
  To evaluate the difference in patient satisfaction associated with FCA exposure (Case v. Control) will be evaluated using chi-square test, t-tests and non-parametric univariate tests distribution dependent. Mean patient and caregiver scores will be calculated for each dyad and compared between groups. Sensitivity analyses may stratify by level of FCA use (low-moderate-high) per dyad and opportunity time for FCA exposure. Case to Control patient analyses will also be performed to detect role-level differences in perceptions of satisfaction associated with FCA exposure.To evaluate the association of the change in patient satisfaction associated with FCA use difference in response between pre- and post- surveys paired t-test or ANCOVA depending on data type and distribution. Within Case Dyads, patient means will be compared with caregiver means to detect difference in satisfaction perceptions based on role.

SECONDARY OUTCOMES:
Caregiver Satisfaction | 8 weeks
  To evaluate the difference in caregiver satisfaction associated with FCA exposure (Case v. Control) will be evaluated using chi-square test, t-tests and non-parametric univariate tests distribution dependent. Mean patient and caregiver scores will be calculated for each dyad and compared between groups. Sensitivity analyses may stratify by level of FCA use (low-moderate-high) per dyad and opportunity time for FCA exposure. Case to Control caregiver analyses will also be performed to detect role-level differences in perceptions of satisfaction associated with FCA exposure. To evaluate the association of the change in caregiver satisfaction associated with FCA use difference in response between pre- and post- surveys paired t-test or ANCOVA depending on data type and distribution. Within Case Dyads, patient means will be compared with caregiver means to detect difference in satisfaction perceptions based on role.
Patient Quality of Life | 8 weeks
  To evaluate the difference in patient quality of life associated with FCA exposure (Case v. Control) will be evaluated using chi-square test, t-tests and non-parametric univariate tests distribution dependent. Mean patient and caregiver scores will be calculated for each dyad and compared between groups. Sensitivity analyses may stratify by level of FCA use (low-moderate-high) per dyad and opportunity time for FCA exposure. Case to Control patient analyses will also be performed to detect role-level differences in perceptions of quality of life associated with FCA exposure.To evaluate the association of the change in patient quality of life associated with FCA use difference in response between pre- and post- surveys paired t-test or ANCOVA depending on data type and distribution. Within Case Dyads, patient means will be compared with caregiver means to detect difference in quality of life perceptions based on role.
Caregiver Quality of Life | 8 weeks
  To evaluate the difference in caregiver quality of life associated with FCA exposure (Case v. Control) will be evaluated using chi-square test, t-tests and non-parametric univariate tests distribution dependent. Mean patient and caregiver scores will be calculated for each dyad and compared between groups. Sensitivity analyses may stratify by level of FCA use (low-moderate-high) per dyad and opportunity time for FCA exposure. Case to Control caregiver analyses will also be performed to detect role-level differences in perceptions of quality of life associated with FCA exposure. To evaluate the association of the change in caregiver quality of life associated with FCA use difference in response between pre- and post- surveys paired t-test or ANCOVA depending on data type and distribution. Within Case Dyads, patient means will be compared with caregiver means to detect difference in quality of life perceptions based on role.
Family Centered Care | 8 weeks
  To evaluate the difference in family centered care associated with FCA exposure (Case v. Control) will be evaluated using chi-square test, t-tests and non-parametric univariate tests distribution dependent. Mean patient and caregiver scores will be calculated for each dyad and compared between groups. Sensitivity analyses may stratify by level of FCA use (low-moderate-high) per dyad and opportunity time for FCA exposure. Case to Control patient and caregiver analyses will also be performed to detect role-level differences in perceptions of family centered care associated with FCA exposure. To evaluate the association of the change in family centered care associated with FCA use difference in response between pre- and post- surveys paired t-test or ANCOVA depending on data type and distribution. Within Case Dyads, patient means will be compared with caregiver means to detect difference in family centered care perceptions based on role.
Patient Experience | 8 weeks
  To evaluate the difference in patient experience associated with FCA exposure (Case v. Control) will be evaluated using chi-square test, t-tests and non-parametric univariate tests distribution dependent. Mean patient and caregiver scores will be calculated for each dyad and compared between groups. Sensitivity analyses may stratify by level of FCA use (low-moderate-high) per dyad and opportunity time for FCA exposure. Case to Control patient analyses will also be performed to detect role-level differences in perceptions of experience associated with FCA exposure.To evaluate the association of the change in patient experience associated with FCA use difference in response between pre- and post- surveys paired t-test or ANCOVA depending on data type and distribution. Within Case Dyads, patient means will be compared with caregiver means to detect difference in experience perceptions based on role.
Caregiver Burden | 8 weeks
  To evaluate the difference in caregiver burden associated with FCA exposure (Case v. Control) will be evaluated using chi-square test, t-tests and non-parametric univariate tests distribution dependent. Mean caregiver scores will be calculated for each dyad and compared between groups. Sensitivity analyses may stratify by level of FCA use (low-moderate-high) per dyad and opportunity time for FCA exposure. Case to Control caregiver analyses will also be performed to detect role-level differences in perceptions of burden associated with FCA exposure.To evaluate the association of the change in caregiver burden associated with FCA use difference in response between pre- and post- surveys paired t-test or ANCOVA depending on data type and distribution. To evaluate the association of the change in caregiver burden associated with FCA use difference in response between pre- and post- surveys paired t-test or ANCOVA depending on data type and distribution.

CONTACTS AND LOCATIONS:
Overall Officials: Lisa Bailey-Davis, DEd, RD, Principal Investigator — Geisinger Clinic
Locations (1):
- Geisinger Health System, Danville, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-05-24): https://cdn.clinicaltrials.gov/large-docs/54/NCT03694054/Prot_SAP_000.pdf